CLINICAL TRIAL: NCT03243396
Title: Building and Sustaining Interventions for Children (BASIC): Task-sharing Mental Health Care in Low-resource Settings
Brief Title: Building and Sustaining Interventions for Children: Task-sharing Mental Health Care in Low-resource Settings
Acronym: BASIC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: University of Washington (Other); Johns Hopkins University (Other); Ace Africa (Other); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: Pro00081913; 1R01MH112633 (NIH)
Record Dates: First submitted 2017-07-13; First posted 2017-08-09 (Actual); Results first posted 2025-04-01 (Actual); Last update posted 2025-04-01 (Actual); Status verified 2025-03

CONDITIONS: Grief; Post Traumatic Stress Disorder; Depression
Keywords: Mental health; Cognitive behavioral therapy; Task-shifting; Global health; Teacher; Community health volunteer; Children; Orphans; Abandoned children; TF-CBT; Mental health policy; Ministry of Education; Ministry of Health; Delivery; Implementation science; Qualitative comparative analysis; Implementation practices and policies; Youth; Adoption; Fidelity; Kenya; Bungoma; Kanduyi; West Africa; Posttraumatic stress; Childhood traumatic grief; Grief; Trauma; Task-sharing; Global mental health
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Depression; Psychological Well-Being; Wounds and Injuries

STUDY DESIGN:
Intervention Model Description: Child mental health outcomes are assessed using an incomplete stepped wedge, cluster randomized controlled trial with 7 sequences. Child participants & one guardian each are randomized to receive the treatment (therapy sessions) from lay counselors in the Health (Community Health Volunteer) or Education (teacher) sector, with timing based on the sequence to which their village cluster was randomly assigned. These participants are the focus of the Interventional Study Design in Aim 3. Also included are lay counselors & site leaders (Head Teachers, Deputy Teachers, & Community Health Extension Workers), given that it is a hybrid effectiveness-implementation trial. These participants, the focus of implementation questions in Aims 1 & 2, provide TF-CBT & do not receive therapy sessions themselves. The village clusters are randomized to sequences in the SW-CRT, & if randomized to sequences 2-7, they receive coaching support informed by sequence 1 on how to effectively implement TF-CBT.
Masking Description: No masking--Child/Adolescent participants and their participating guardian will be able to tell to which arm they were allocated or randomized, given that they know from whom they receive treatment (from teachers, indicating Education or from Community Health Volunteers, indicating Health). There are other participant types in addition to children/adolescents and guardians who are enrolled in BASIC (per above description) to answer implementation questions (Aims 1 and 2 of BASIC). As noted above, these other participants include the lay counselors (teachers and Community Health Volunteers, their site leaders [Education: Head Teachers and Deputy Teachers; Health: Community Health Extension Workers]).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Health-Sector Delivered CBT (Experimental): These child/adolescent participants and one of their guardians will receive Pamoja Tunaweza, the locally adapted version of Trauma-Focused Cognitive Behavioral Therapy, in a community setting from Community Health Volunteers.
  Interventions: Behavioral: Trauma-Focused Cognitive Behavioral Therapy
- Education-Sector Delivered CBT (Experimental): These child/adolescent participants and one of their guardians will receive Pamoja Tunaweza, the locally adapted version of Trauma-Focused Cognitive Behavioral Therapy, in their school setting from teachers employed by their school.
  Interventions: Behavioral: Trauma-Focused Cognitive Behavioral Therapy

INTERVENTIONS:
Behavioral: Trauma-Focused Cognitive Behavioral Therapy — Eight small-group sessions, including eight children and one guardian for each child, will meet separately, with joint activities in the final three sessions. TF-CBT will be delivered via community health volunteers in the community setting, and via selected teachers in the school setting--with two lay counselors leading the child group, and one leading the guardian group. Most TF-CBT components (psychoeducation, parenting, relaxation, cognitive coping, grief specific skills) will be delivered in groups, but 2-3 individual sessions mid-group will be used for imaginal exposure (i.e., talking about/processing traumatic events).
  Other Names: Pamoja Tunaweza

SUMMARY:
The BASIC study will take place in Kanduyi/Bungoma South Sub-County, in western Kenya, and focuses on children orphaned by one or two parents. Growing evidence demonstrates that orphaned children in low- and middle-income countries are at higher risk of mental health problems, but mental health professionals are largely unavailable in this area. Research suggests that some mental health treatments can be delivered effectively in low- and middle-income countries using a task-shifting approach, in which lay counselors with little or no prior mental health experience are trained to provide treatment, and deliver with supervision. However, very little is known about how to support local systems and organizations in delivering mental health care via task-shifting, particularly in a way that could scale-able and sustainable in the low-resource context. The BASIC team's prior work suggests that partnering with two government sectors, education and health, could be a low-cost and sustainable strategy to implement task-shifted mental health services. By training teachers (via the Education sector) and community health volunteers (via the Health sector) to provide mental health care, a larger population could potentially be reached. Before attempting any country or system-wide implementation, it is important to know what is needed to enable successful implementation in either or both sectors, client outcomes for those receiving mental health care when delivered via Education or Health, and cost of delivery in both sectors. The team aims to collect outcomes that are relevant to policy makers, and that can be considered along with cost and experiences in both sectors.

DETAILED DESCRIPTION:
Building and Sustaining Interventions for Children (BASIC): Task-sharing mental health care in low-resource settings builds on our 15-year history of collaborations with research partners in Kenya, prior NIH-funded work that identified mental health needs of orphaned children in low- and middle-income countries, and iterative and collaborative intervention adaptation and testing using a task-sharing approach, to address these needs.Our goal is to identify locally sustainable implementation policies and practices (IPPs) that lead to effective implementation of task-shared evidence-based treatment (EBT) delivery (a locally adapted version of Trauma-focused Cognitive Behavioral Therapy (TF-CBT), Pamoja Tunaweza in this study) in 2 governmental sectors in Kenya. Both sectors were identified by our Kenyan partners as potential platforms for scale- up-Education via teacher delivery and Health via community health volunteer (CHV) delivery. Both Education and Health may be viable sectors for mental health care delivery, but the IPPs that predict implementation success and intervention effectiveness in either/ both sectors are unknown. This study identifies con-textually relevant, practical, and actionable IPPs that can inform implementation planning, while also assessing child outcomes and intervention costs in both sectors.

The recent devolvement of the Kenyan government (leading to more local decision-making), the launch of a National Mental Health Policy, and our Kenyan partners' empowerment work building enthusiasm for TF-CBT are converging to create a local climate in which BASIC could become part of the county plan, if evidence-based guidance for implementation, using mostly existing resources, existed. The trial design is an incomplete stepped wedge cluster randomized controlled trial (SW-CRT) including 40 schools and the 40 surrounding villages. The school and the surrounding community are considered a "village cluster." Each of the 40 "village clusters" has 1 team of teachers and 1 team of CHVs delivering Pamoja Tunaweza, resulting in 120 trained lay counselors in each sector, who provide TF-CBT to 1,280 youth and one of their guardians, across seven sequences of the SW-CRT. Site leaders are enrolled for data collection (up to 80), but do not provide services. The study uses a novel method, qualitative comparative analyses (QCA), that holds potential for substantially advancing the field of implementation science. QCA leverages the rigor of quantitative approaches and the detail of qualitative approaches, and allows for complex causality and equifinality (i.e., an outcome can be reached by multiple means).

Study aims are: 1) Identify actionable IPPs that predict adoption (delivery) and fidelity (high- quality delivery) after 10 sites in each sector implement TF-CBT (sequence 1). Use identified IPPs to (Aim 1a) guide implementation planning support for subsequent sites and to (Aim 1b) generate testable hypotheses about IPPs as causal mechanisms; 2) Test mechanisms of implementation success in both sectors across all 7 sequences; and 3) Test TF-CBT effectiveness (i.e., mental health outcomes; functioning) and cost in both sectors. This research has important implications for implementing an evidence-based treatment in low-resource settings, including the US.

ELIGIBILITY:
Inclusion Criteria:

* Child or young adolescent between the ages of 11 and 14 at the time of enrollment
* Child lost one or both parents to death at least 6 months ago or later, and when the child was 4 years old or older
* Child lives in the community with at least one adult guardian (18 years old or older)
* Child is experiencing borderline or clinically significant levels of post-traumatic stress or childhood traumatic grief (as indicated by a score of 18 or higher on the Child Posttraumatic Stress Scale, or a score of 35 or higher on the Inventory of Complicated Grief)

Exclusion Criteria:

* Child has a known developmental or cognitive disability
* Child attends private school
* Child and family are about to move
* Children who lost a parent less than 6 months ago (since they may be experiencing a normal grief reaction and may not necessarily be in need of the treatment for CTG)
* Caregiver of the child refuses to participate
* Lay counselor is not literate
* Lay counselor does not have a mobile phone
* Lay counselor refuses to serve as a counselor
* Site leader refuses to allow their site to participate in the study

Ages: 11 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 956 (Actual)
Dates: Start 2018-02-01 (Actual); Primary Completion 2024-01-25 (Actual); Study Completion 2024-01-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kathryn Whetten, PhD, Principal Investigator — Center for Health Policy and Inequalities Research at Duke University; Shannon Dorsey, PhD, Principal Investigator — University of Washington Department of Psychology
Locations (1):
- ACE Africa, Bungoma, Bungoma County, Kenya

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Thornicroft G, Alem A, Antunes Dos Santos R, Barley E, Drake RE, Gregorio G, Hanlon C, Ito H, Latimer E, Law A, Mari J, McGeorge P, Padmavati R, Razzouk D, Semrau M, Setoya Y, Thara R, Wondimagegn D. WPA guidance on steps, obstacles and mistakes to avoid in the implementation of community mental health care. World Psychiatry. 2010 Jun;9(2):67-77. doi: 10.1002/j.2051-5545.2010.tb00276.x. PMID 20671888
- [Background] Saxena S, Thornicroft G, Knapp M, Whiteford H. Resources for mental health: scarcity, inequity, and inefficiency. Lancet. 2007 Sep 8;370(9590):878-89. doi: 10.1016/S0140-6736(07)61239-2. PMID 17804062
- [Background] Eaton J, McCay L, Semrau M, Chatterjee S, Baingana F, Araya R, Ntulo C, Thornicroft G, Saxena S. Scale up of services for mental health in low-income and middle-income countries. Lancet. 2011 Oct 29;378(9802):1592-603. doi: 10.1016/S0140-6736(11)60891-X. Epub 2011 Oct 16. PMID 22008429
- [Background] Betancourt TS, Chambers DA. Optimizing an Era of Global Mental Health Implementation Science. JAMA Psychiatry. 2016 Feb;73(2):99-100. doi: 10.1001/jamapsychiatry.2015.2705. No abstract available. PMID 26720304
- [Background] Patel V, Chowdhary N, Rahman A, Verdeli H. Improving access to psychological treatments: lessons from developing countries. Behav Res Ther. 2011 Sep;49(9):523-8. doi: 10.1016/j.brat.2011.06.012. Epub 2011 Jul 7. PMID 21788012
- [Background] Cragun D, Radford C, Dolinsky JS, Caldwell M, Chao E, Pal T. Panel-based testing for inherited colorectal cancer: a descriptive study of clinical testing performed by a US laboratory. Clin Genet. 2014 Dec;86(6):510-20. doi: 10.1111/cge.12359. Epub 2014 Mar 20. PMID 24506336
- [Background] McAlearney AS, Walker D, Moss AD, Bickell NA. Using Qualitative Comparative Analysis of Key Informant Interviews in Health Services Research: Enhancing a Study of Adjuvant Therapy Use in Breast Cancer Care. Med Care. 2016 Apr;54(4):400-5. doi: 10.1097/MLR.0000000000000503. PMID 26908085
- [Background] Marcus Thygeson N, Solberg LI, Asche SE, Fontaine P, Gregory Pawlson L, Scholle SH. Using fuzzy set qualitative comparative analysis (fs/QCA) to explore the relationship between medical "homeness" and quality. Health Serv Res. 2012 Feb;47(1 Pt 1):22-45. doi: 10.1111/j.1475-6773.2011.01303.x. Epub 2011 Aug 22. PMID 22092269
- [Background] Curran GM, Bauer M, Mittman B, Pyne JM, Stetler C. Effectiveness-implementation hybrid designs: combining elements of clinical effectiveness and implementation research to enhance public health impact. Med Care. 2012 Mar;50(3):217-26. doi: 10.1097/MLR.0b013e3182408812. PMID 22310560
- [Background] Kohn R, Saxena S, Levav I, Saraceno B. The treatment gap in mental health care. Bull World Health Organ. 2004 Nov;82(11):858-66. Epub 2004 Dec 14. PMID 15640922
- [Background] Thornicroft G, Cooper S, Bortel TV, Kakuma R, Lund C. Capacity building in global mental health research. Harv Rev Psychiatry. 2012 Jan-Feb;20(1):13-24. doi: 10.3109/10673229.2012.649117. PMID 22335179
- [Background] Patel V. The future of psychiatry in low- and middle-income countries. Psychol Med. 2009 Nov;39(11):1759-62. doi: 10.1017/s0033291709005224. PMID 20162837
- [Background] Patel V, Araya R, Chatterjee S, Chisholm D, Cohen A, De Silva M, Hosman C, McGuire H, Rojas G, van Ommeren M. Treatment and prevention of mental disorders in low-income and middle-income countries. Lancet. 2007 Sep 15;370(9591):991-1005. doi: 10.1016/S0140-6736(07)61240-9. PMID 17804058
- [Background] van Ginneken N, Tharyan P, Lewin S, Rao GN, Meera SM, Pian J, Chandrashekar S, Patel V. Non-specialist health worker interventions for the care of mental, neurological and substance-abuse disorders in low- and middle-income countries. Cochrane Database Syst Rev. 2013 Nov 19;(11):CD009149. doi: 10.1002/14651858.CD009149.pub2. PMID 24249541
- [Background] Bolton P, Bass J, Neugebauer R, Verdeli H, Clougherty KF, Wickramaratne P, Speelman L, Ndogoni L, Weissman M. Group interpersonal psychotherapy for depression in rural Uganda: a randomized controlled trial. JAMA. 2003 Jun 18;289(23):3117-24. doi: 10.1001/jama.289.23.3117. PMID 12813117
- [Background] Bolton P, Bass J, Betancourt T, Speelman L, Onyango G, Clougherty KF, Neugebauer R, Murray L, Verdeli H. Interventions for depression symptoms among adolescent survivors of war and displacement in northern Uganda: a randomized controlled trial. JAMA. 2007 Aug 1;298(5):519-27. doi: 10.1001/jama.298.5.519. PMID 17666672
- [Background] Patel V, Weiss HA, Chowdhary N, Naik S, Pednekar S, Chatterjee S, De Silva MJ, Bhat B, Araya R, King M, Simon G, Verdeli H, Kirkwood BR. Effectiveness of an intervention led by lay health counsellors for depressive and anxiety disorders in primary care in Goa, India (MANAS): a cluster randomised controlled trial. Lancet. 2010 Dec 18;376(9758):2086-95. doi: 10.1016/S0140-6736(10)61508-5. Epub 2010 Dec 13. PMID 21159375
- [Background] Weiss WM, Murray LK, Zangana GA, Mahmooth Z, Kaysen D, Dorsey S, Lindgren K, Gross A, Murray SM, Bass JK, Bolton P. Community-based mental health treatments for survivors of torture and militant attacks in Southern Iraq: a randomized control trial. BMC Psychiatry. 2015 Oct 14;15:249. doi: 10.1186/s12888-015-0622-7. PMID 26467303
- [Background] Murray LK, Skavenski S, Kane JC, Mayeya J, Dorsey S, Cohen JA, Michalopoulos LT, Imasiku M, Bolton PA. Effectiveness of Trauma-Focused Cognitive Behavioral Therapy Among Trauma-Affected Children in Lusaka, Zambia: A Randomized Clinical Trial. JAMA Pediatr. 2015 Aug;169(8):761-9. doi: 10.1001/jamapediatrics.2015.0580. PMID 26111066
- [Background] McMullen J, O'Callaghan P, Shannon C, Black A, Eakin J. Group trauma-focused cognitive-behavioural therapy with former child soldiers and other war-affected boys in the DR Congo: a randomised controlled trial. J Child Psychol Psychiatry. 2013 Nov;54(11):1231-41. doi: 10.1111/jcpp.12094. Epub 2013 Jun 6. PMID 23738530
- [Background] O'Callaghan P, McMullen J, Shannon C, Rafferty H, Black A. A randomized controlled trial of trauma-focused cognitive behavioral therapy for sexually exploited, war-affected Congolese girls. J Am Acad Child Adolesc Psychiatry. 2013 Apr;52(4):359-69. doi: 10.1016/j.jaac.2013.01.013. Epub 2013 Mar 6. PMID 23582867
- [Background] Rahman A, Malik A, Sikander S, Roberts C, Creed F. Cognitive behaviour therapy-based intervention by community health workers for mothers with depression and their infants in rural Pakistan: a cluster-randomised controlled trial. Lancet. 2008 Sep 13;372(9642):902-9. doi: 10.1016/S0140-6736(08)61400-2. PMID 18790313
- [Background] Bass J, Neugebauer R, Clougherty KF, Verdeli H, Wickramaratne P, Ndogoni L, Speelman L, Weissman M, Bolton P. Group interpersonal psychotherapy for depression in rural Uganda: 6-month outcomes: randomised controlled trial. Br J Psychiatry. 2006 Jun;188:567-73. doi: 10.1192/bjp.188.6.567. PMID 16738348
- [Background] Murray LK, Skavenski S, Michalopoulos LM, Bolton PA, Bass JK, Familiar I, Imasiku M, Cohen J. Counselor and client perspectives of Trauma-focused Cognitive Behavioral Therapy for children in Zambia: a qualitative study. J Clin Child Adolesc Psychol. 2014;43(6):902-14. doi: 10.1080/15374416.2013.859079. Epub 2014 Jan 8. PMID 24400677
- [Background] Hanlon C, Luitel NP, Kathree T, Murhar V, Shrivasta S, Medhin G, Ssebunnya J, Fekadu A, Shidhaye R, Petersen I, Jordans M, Kigozi F, Thornicroft G, Patel V, Tomlinson M, Lund C, Breuer E, De Silva M, Prince M. Challenges and opportunities for implementing integrated mental health care: a district level situation analysis from five low- and middle-income countries. PLoS One. 2014 Feb 18;9(2):e88437. doi: 10.1371/journal.pone.0088437. eCollection 2014. PMID 24558389
- [Background] Glasgow RE, Fisher L, Strycker LA, Hessler D, Toobert DJ, King DK, Jacobs T. Minimal intervention needed for change: definition, use, and value for improving health and health research. Transl Behav Med. 2014 Mar;4(1):26-33. doi: 10.1007/s13142-013-0232-1. PMID 24653774
- [Background] McClure JB, Derry H, Riggs KR, Westbrook EW, St John J, Shortreed SM, Bogart A, An LC. Questions about quitting (Q2): design and methods of a Multiphase Optimization Strategy (MOST) randomized screening experiment for an online, motivational smoking cessation intervention. Contemp Clin Trials. 2012 Sep;33(5):1094-102. doi: 10.1016/j.cct.2012.06.009. Epub 2012 Jul 4. PMID 22771577
- [Background] Iwelunmor J, Blackstone S, Veira D, Nwaozuru U, Airhihenbuwa C, Munodawafa D, Kalipeni E, Jutal A, Shelley D, Ogedegebe G. Toward the sustainability of health interventions implemented in sub-Saharan Africa: a systematic review and conceptual framework. Implement Sci. 2016 Mar 23;11:43. doi: 10.1186/s13012-016-0392-8. PMID 27005280
- [Background] Chambers DA, Glasgow RE, Stange KC. The dynamic sustainability framework: addressing the paradox of sustainment amid ongoing change. Implement Sci. 2013 Oct 2;8:117. doi: 10.1186/1748-5908-8-117. PMID 24088228
- [Background] Ghiron L, Shillingi L, Kabiswa C, Ogonda G, Omimo A, Ntabona A, Simmons R, Fajans P. Beginning with sustainable scale up in mind: initial results from a population, health and environment project in East Africa. Reprod Health Matters. 2014 May;22(43):84-92. doi: 10.1016/S0968-8080(14)43761-3. PMID 24908459
- [Background] Sherr K, Gimbel S, Rustagi A, Nduati R, Cuembelo F, Farquhar C, Wasserheit J, Gloyd S; With input from the SAIA Study Team. Systems analysis and improvement to optimize pMTCT (SAIA): a cluster randomized trial. Implement Sci. 2014 May 8;9:55. doi: 10.1186/1748-5908-9-55. PMID 24885976
- [Background] Shelley D, VanDevanter N, Cleland CC, Nguyen L, Nguyen N. Implementing tobacco use treatment guidelines in community health centers in Vietnam. Implement Sci. 2015 Oct 9;10:142. doi: 10.1186/s13012-015-0328-8. PMID 26453554
- [Background] Whetten K, Ostermann J, Whetten R, O'Donnell K, Thielman N; Positive Outcomes for Orphans Research Team. More than the loss of a parent: potentially traumatic events among orphaned and abandoned children. J Trauma Stress. 2011 Apr;24(2):174-82. doi: 10.1002/jts.20625. Epub 2011 Mar 25. PMID 21442663
- [Background] Gray CL, Pence BW, Ostermann J, Whetten RA, O'Donnell K, Thielman NM, Whetten K. Gender (in) differences in prevalence and incidence of traumatic experiences among orphaned and separated children living in five low- and middle-income countries. Glob Ment Health (Camb). 2015 Jan;2:e3. doi: 10.1017/gmh.2015.1. PMID 26085939
- [Background] Thielman N, Ostermann J, Whetten K, Whetten R, O'Donnell K; Positive Outcomes for Orphans Research Team. Correlates of poor health among orphans and abandoned children in less wealthy countries: the importance of caregiver health. PLoS One. 2012;7(6):e38109. doi: 10.1371/journal.pone.0038109. Epub 2012 Jun 13. PMID 22719867
- [Background] Escueta M, Whetten K, Ostermann J, O'Donnell K; Positive Outcomes for Orphans Research Team. Adverse childhood experiences, psychosocial well-being and cognitive development among orphans and abandoned children in five low income countries. BMC Int Health Hum Rights. 2014 Mar 10;14:6. doi: 10.1186/1472-698X-14-6. PMID 24606949
- [Background] Hemming K, Haines TP, Chilton PJ, Girling AJ, Lilford RJ. The stepped wedge cluster randomised trial: rationale, design, analysis, and reporting. BMJ. 2015 Feb 6;350:h391. doi: 10.1136/bmj.h391. No abstract available. PMID 25662947
- [Background] mhGAP Intervention Guide for Mental, Neurological and Substance Use Disorders in Non-Specialized Health Settings: Mental Health Gap Action Programme (mhGAP). Geneva: World Health Organization; 2010. Available from http://www.ncbi.nlm.nih.gov/books/NBK138690/ PMID 23741783
- [Background] Saldana L, Chamberlain P. Supporting implementation: the role of community development teams to build infrastructure. Am J Community Psychol. 2012 Dec;50(3-4):334-46. doi: 10.1007/s10464-012-9503-0. PMID 22430709
- [Background] Hurlburt M, Aarons GA, Fettes D, Willging C, Gunderson L, Chaffin MJ. Interagency Collaborative Team Model for Capacity Building to Scale-Up Evidence-Based Practice. Child Youth Serv Rev. 2014 Apr;39:160-168. doi: 10.1016/j.childyouth.2013.10.005. PMID 27512239
- [Background] Kiima D, Jenkins R. Mental health policy in Kenya -an integrated approach to scaling up equitable care for poor populations. Int J Ment Health Syst. 2010 Jun 28;4:19. doi: 10.1186/1752-4458-4-19. PMID 20584266
- [Background] Takasugi T, Lee AC. Why do community health workers volunteer? A qualitative study in Kenya. Public Health. 2012 Oct;126(10):839-45. doi: 10.1016/j.puhe.2012.06.005. Epub 2012 Oct 1. PMID 23036777
- [Background] Weiner BJ, Lewis MA, Linnan LA. Using organization theory to understand the determinants of effective implementation of worksite health promotion programs. Health Educ Res. 2009 Apr;24(2):292-305. doi: 10.1093/her/cyn019. Epub 2008 May 9. PMID 18469319
- [Background] Silverman WK, Ortiz CD, Viswesvaran C, Burns BJ, Kolko DJ, Putnam FW, Amaya-Jackson L. Evidence-based psychosocial treatments for children and adolescents exposed to traumatic events. J Clin Child Adolesc Psychol. 2008 Jan;37(1):156-83. doi: 10.1080/15374410701818293. PMID 18444057
- [Background] Dorsey S, McLaughlin KA, Kerns SEU, Harrison JP, Lambert HK, Briggs EC, Revillion Cox J, Amaya-Jackson L. Evidence Base Update for Psychosocial Treatments for Children and Adolescents Exposed to Traumatic Events. J Clin Child Adolesc Psychol. 2017 May-Jun;46(3):303-330. doi: 10.1080/15374416.2016.1220309. Epub 2016 Oct 19. PMID 27759442
- [Background] Dorsey S, Pullmann MD, Berliner L, Koschmann E, McKay M, Deblinger E. Engaging foster parents in treatment: a randomized trial of supplementing trauma-focused cognitive behavioral therapy with evidence-based engagement strategies. Child Abuse Negl. 2014 Sep;38(9):1508-20. doi: 10.1016/j.chiabu.2014.03.020. Epub 2014 Apr 29. PMID 24791605
- [Background] O'Donnell K, Dorsey S, Gong W, Ostermann J, Whetten R, Cohen JA, Itemba D, Manongi R, Whetten K. Treating maladaptive grief and posttraumatic stress symptoms in orphaned children in Tanzania: group-based trauma-focused cognitive-behavioral therapy. J Trauma Stress. 2014 Dec;27(6):664-71. doi: 10.1002/jts.21970. Epub 2014 Nov 21. PMID 25418514
- [Background] Deblinger E, Pollio E, Dorsey S. Applying Trauma-Focused Cognitive-Behavioral Therapy in Group Format. Child Maltreat. 2016 Feb;21(1):59-73. doi: 10.1177/1077559515620668. Epub 2015 Dec 23. PMID 26701151
- [Background] Woods-Jaeger BA, Kava CM, Akiba CF, Lucid L, Dorsey S. The art and skill of delivering culturally responsive trauma-focused cognitive behavioral therapy in Tanzania and Kenya. Psychol Trauma. 2017 Mar;9(2):230-238. doi: 10.1037/tra0000170. Epub 2016 Jul 14. PMID 27414470
- [Background] Beidas RS, Kendall PC. Training Therapists in Evidence-Based Practice: A Critical Review of Studies From a Systems-Contextual Perspective. Clin Psychol (New York). 2010 Mar;17(1):1-30. doi: 10.1111/j.1468-2850.2009.01187.x. PMID 20877441
- [Background] Chamberlain P, Price J, Reid J, Landsverk J. Cascading implementation of a foster and kinship parent intervention. Child Welfare. 2008;87(5):27-48. PMID 19402358
- [Background] Herschell AD, Kolko DJ, Baumann BL, Davis AC. The role of therapist training in the implementation of psychosocial treatments: a review and critique with recommendations. Clin Psychol Rev. 2010 Jun;30(4):448-66. doi: 10.1016/j.cpr.2010.02.005. Epub 2010 Mar 1. PMID 20304542
- [Background] Leontjevas R, Gerritsen DL, Smalbrugge M, Teerenstra S, Vernooij-Dassen MJ, Koopmans RT. A structural multidisciplinary approach to depression management in nursing-home residents: a multicentre, stepped-wedge cluster-randomised trial. Lancet. 2013 Jun 29;381(9885):2255-64. doi: 10.1016/S0140-6736(13)60590-5. Epub 2013 May 2. PMID 23643110
- [Background] Murray LK, Dorsey S, Bolton P, Jordans MJ, Rahman A, Bass J, Verdeli H. Building capacity in mental health interventions in low resource countries: an apprenticeship model for training local providers. Int J Ment Health Syst. 2011 Nov 18;5(1):30. doi: 10.1186/1752-4458-5-30. PMID 22099582
- [Background] Kane H, Lewis MA, Williams PA, Kahwati LC. Using qualitative comparative analysis to understand and quantify translation and implementation. Transl Behav Med. 2014 Jun;4(2):201-8. doi: 10.1007/s13142-014-0251-6. PMID 24904704
- [Background] Weiner BJ, Jacobs SR, Minasian LM, Good MJ. Organizational designs for achieving high treatment trial enrollment: a fuzzy-set analysis of the community clinical oncology program. J Oncol Pract. 2012 Sep;8(5):287-91. doi: 10.1200/JOP.2011.000507. Epub 2012 May 1. PMID 23277765
- [Background] Proctor E, Silmere H, Raghavan R, Hovmand P, Aarons G, Bunger A, Griffey R, Hensley M. Outcomes for implementation research: conceptual distinctions, measurement challenges, and research agenda. Adm Policy Ment Health. 2011 Mar;38(2):65-76. doi: 10.1007/s10488-010-0319-7. PMID 20957426
- [Background] Damschroder LJ, Aron DC, Keith RE, Kirsh SR, Alexander JA, Lowery JC. Fostering implementation of health services research findings into practice: a consolidated framework for advancing implementation science. Implement Sci. 2009 Aug 7;4:50. doi: 10.1186/1748-5908-4-50. PMID 19664226
- [Background] Glasgow RE, Vogt TM, Boles SM. Evaluating the public health impact of health promotion interventions: the RE-AIM framework. Am J Public Health. 1999 Sep;89(9):1322-7. doi: 10.2105/ajph.89.9.1322. PMID 10474547
- [Background] Luke DA, Calhoun A, Robichaux CB, Elliott MB, Moreland-Russell S. The Program Sustainability Assessment Tool: a new instrument for public health programs. Prev Chronic Dis. 2014 Jan 23;11:130184. doi: 10.5888/pcd11.130184. PMID 24456645
- [Background] Baker R, Camosso-Stefinovic J, Gillies C, Shaw EJ, Cheater F, Flottorp S, Robertson N, Wensing M, Fiander M, Eccles MP, Godycki-Cwirko M, van Lieshout J, Jager C. Tailored interventions to address determinants of practice. Cochrane Database Syst Rev. 2015 Apr 29;2015(4):CD005470. doi: 10.1002/14651858.CD005470.pub3. PMID 25923419
- [Background] Baker R, Camosso-Stefinovic J, Gillies C, Shaw EJ, Cheater F, Flottorp S, Robertson N. Tailored interventions to overcome identified barriers to change: effects on professional practice and health care outcomes. Cochrane Database Syst Rev. 2010 Mar 17;(3):CD005470. doi: 10.1002/14651858.CD005470.pub2. PMID 20238340
- [Background] Powell BJ, Beidas RS, Lewis CC, Aarons GA, McMillen JC, Proctor EK, Mandell DS. Methods to Improve the Selection and Tailoring of Implementation Strategies. J Behav Health Serv Res. 2017 Apr;44(2):177-194. doi: 10.1007/s11414-015-9475-6. PMID 26289563
- [Background] Bosch M, van der Weijden T, Wensing M, Grol R. Tailoring quality improvement interventions to identified barriers: a multiple case analysis. J Eval Clin Pract. 2007 Apr;13(2):161-8. doi: 10.1111/j.1365-2753.2006.00660.x. PMID 17378860
- [Background] Wiltsey Stirman S, Kimberly J, Cook N, Calloway A, Castro F, Charns M. The sustainability of new programs and innovations: a review of the empirical literature and recommendations for future research. Implement Sci. 2012 Mar 14;7:17. doi: 10.1186/1748-5908-7-17. PMID 22417162
- [Background] Whelan J, Love P, Pettman T, Doyle J, Booth S, Smith E, Waters E. Cochrane update: Predicting sustainability of intervention effects in public health evidence: identifying key elements to provide guidance. J Public Health (Oxf). 2014 Jun;36(2):347-51. doi: 10.1093/pubmed/fdu027. Epub 2014 May 23. No abstract available. PMID 24860152
- [Background] Dorsey S, Lucid L, Murray L, Bolton P, Itemba D, Manongi R, Whetten K. A Qualitative Study of Mental Health Problems Among Orphaned Children and Adolescents in Tanzania. J Nerv Ment Dis. 2015 Nov;203(11):864-70. doi: 10.1097/NMD.0000000000000388. PMID 26488916
- [Background] Hussey MA, Hughes JP. Design and analysis of stepped wedge cluster randomized trials. Contemp Clin Trials. 2007 Feb;28(2):182-91. doi: 10.1016/j.cct.2006.05.007. Epub 2006 Jul 7. PMID 16829207
- [Background] Seaman SR, White IR. Review of inverse probability weighting for dealing with missing data. Stat Methods Med Res. 2013 Jun;22(3):278-95. doi: 10.1177/0962280210395740. Epub 2011 Jan 10. PMID 21220355
- [Background] Seaman SR, White IR, Copas AJ, Li L. Combining multiple imputation and inverse-probability weighting. Biometrics. 2012 Mar;68(1):129-37. doi: 10.1111/j.1541-0420.2011.01666.x. Epub 2011 Nov 3. PMID 22050039
- [Background] Seaman SR, Bartlett JW, White IR. Multiple imputation of missing covariates with non-linear effects and interactions: an evaluation of statistical methods. BMC Med Res Methodol. 2012 Apr 10;12:46. doi: 10.1186/1471-2288-12-46. PMID 22489953
- [Background] Hemming K, Taljaard M. Sample size calculations for stepped wedge and cluster randomised trials: a unified approach. J Clin Epidemiol. 2016 Jan;69:137-46. doi: 10.1016/j.jclinepi.2015.08.015. Epub 2015 Sep 5. PMID 26344808
- [Background] Girling AJ, Hemming K. Statistical efficiency and optimal design for stepped cluster studies under linear mixed effects models. Stat Med. 2016 Jun 15;35(13):2149-66. doi: 10.1002/sim.6850. Epub 2016 Jan 7. PMID 26748662
- [Background] Dranove D. Measuring cost. In: Sloan F, ed. Valuing Health Care: Costs, Benefits and Effectiveness. Cambridge University Press; 1995.
- [Background] Haddix AC, Teutsch SM, Corso PS, eds. Prevention Effectiveness: A Guide to Decision Analysis and Economic Evaluation. 2nd ed. Oxford University Press; 2002.
- [Background] Little R, Rubin D. Statistical Analysis with Missing Data. New York: Wiley; 2002.
- [Background] World Health Organization. Beginning with the end in mind: planning pilot projects and other programmatic research for successful scaling up. http://www.who.int/reproductivehealth/publications/strategic_approach/9789241502320/en/. Accessed May 24, 2016.
- [Background] Yin RK. Case Study Research: Design and Methods. Vol 5. Thousand Oaks, CA: SAGE Publications, Inc.; 2009.
- [Background] Trochim WMK. Research Methods Knowledge Base. 2nd ed. Mason, OH: Atomic Dog Publishing; 2001.
- [Background] Miles MB, Huberman AM. Qualitative Data Analysis: An Expanded Sourcebook. SAGE; 1994.
- [Background] Yin RK. Changing Urban Bureaucracies: How New Practices Become Routinized. Lexington, MA: Lexington Books; 1979.
- [Background] Brownson RC, Colditz GA, Proctor EK, eds. Dissemination and Implementation Research in Health: Translating Science to Practice. 1st ed. Oxford, UK: Oxford University Press; 2012.
- [Background] Beebe J. Rapid Qualitative Inquiry: A Field Guide to Team-Based Assessment. 2nd ed. Lanham, Maryland: Rowman & Littlefield; 2014.
- [Background] Jacobs SR, Weiner BJ, Minasian LM, Good MJ. Achieving high cancer control trial enrollment in the community setting: an analysis of the Community Clinical Oncology Program. Contemp Clin Trials. 2013 Mar;34(2):320-5. doi: 10.1016/j.cct.2012.12.008. Epub 2013 Jan 5. PMID 23295315
- [Background] Belden CM, Weiner BJ. A fuzzy set analysis of implementation strategies promoting minority participation in cancer clinical trials. under review.
- [Background] Ferlie E, Fitzgerald L, Wood M, Hawkins C. The Nonspread of Innovations: The Mediating Role of Professionals. The Academy of Management Journal. 2005;48(1):117-134. doi:10.2307/20159644.
- [Background] Van de Ven AH, Polley DE, Garud R, Venkataraman S. The Innovation Journey.; 1999. http://library.wur.nl/WebQuery/clc/1882056. Accessed May 9, 2016.
- [Background] Goertz G, Mahoney J. Two-level theories and fuzzy-set analysis. Sociological Methods & Research. 2005;33(4):497-538. doi:10.1177/0049124104266128.
- [Background] Longest KC, Thoits PA. Gender, the stress process, and health: A configurational approach. Society and Mental Health. 2012;2(3):187-206. doi:10.1177/2156869312451151.
- [Background] Ragin CC. Fuzzy-Set Social Science. University of Chicago Press; 2000.
- [Background] Ragin CC. Redesigning Social Inquiry: Fuzzy Sets and Beyond. University of Chicago Press Chicago; 2008.
- [Background] Avdagic S. When are concerted reforms feasible? Explaining the emergence of social pacts in Western Europe. Comparative Political Studies. 2010;42:628-657.
- [Background] Weiner DA, Schneider A, Lyons JS. Evidence-based treatments for trauma among culturally diverse foster care youth: Treatment retention and outcomes. Children and Youth Services Review. 2009;31:1199- 1205.
- [Background] Ford JK, Weissbein DA. Transfer of training: An updated review and analysis. Performance Improvement Quarterly. 1997;10(2):22-41.
- [Background] Blume BD, Ford JK, Baldwin TT, Huang JL. Transfer of training: A meta-analytic Review. Journal of Management. 2010;36(4):1065-1105.
- [Background] Baldwin TT, Ford JK. Transfer of training: A review and directions for future research. Personnel Psychology. 1988;41(1):63-105.
- [Background] UNICEF. Primary School Years: The Children - Kenya. http://www.unicef.org/kenya/children_3795.htm. Accessed May 25, 2016.
- [Background] World Bank. Data: Population, ages 0-14 (% of total). http://data.worldbank.org/indicator/SP.POP.0014.TO.ZS. Accessed May 25, 2016.
- [Background] Index Mundi. Kenya Demographics Profile 2014. http://www.indexmundi.com/kenya/demographics_profile.html. Accessed May 26, 2016.
- [Background] Ministry of Medical Services, Republic of Kenya. The Mental Health Report. 2nd Draft. Nairobi, Kenya; 2012.
- [Background] Kenyan National Assembly. Mental Health Bill.; 2014.
- [Background] World Bank. Kenya's Devolution. http://www.worldbank.org/en/country/kenya/brief/kenyas-devolution. Accessed May 25, 2016.
- [Background] National Council for Law Reporting (Kenya Law). Kenya Law: Laws on Devolution. Kenya Law. http://kenyalaw.org/kl/index.php?id=3979. Accessed May 25, 2016.
- [Background] UNICEF. Kenya Statistics. http://www.unicef.org/infobycountry/kenya_statistics.html. Accessed April 24, 2016.
- [Background] UNICEF. State of the World's Children: Statistical Tables.; 2015.
- [Background] UNICEF. Africa's Orphaned and Vulnerable Generations: Children Affected by AIDS. Author; 2006. 5/25/2016.
- [Background] Orphans. UNICEF. http://www.unicef.org/media/media_45279.html. Accessed May 25, 2016.
- [Background] Institute of Medicines of the National Academies. Evaluation of PEPFAR. Washington, D.C.: National Academies Press; 2013. http://www.nap.edu/catalog/18256. Accessed May 25, 2016.
- [Background] Muraya J. Kenya Turns Attention to Mental Health With New Policy. AllAfrica. http://allafrica.com/stories/201605181158.html. Published May 18, 2016. Accessed May 30, 2016.
- [Background] World Health Organization. Mental Health Action Plan: 2013-2020. Geneva, Switzerland: Author; 2013.
- [Background] Fairall L, Zwarenstein M, Thornicroft G. The applicability of trials of complex mental health interventions. In: Thornicroft G, Patel V, eds. Global Mental Health Trials. Oxford, UK: Oxford University Press; 2014.
- [Background] World Health Organization. Mental Health Atlas 2011. 2011. http://www.who.int/mental_health/publications/mental_health_atlas_2011/en/.
- [Background] World Health Organization. Global Burden of Disease Report: 2004 Update. Geneva, Switzerland: Author; 2008.
- [Derived] Triplett NS, Munson S, Mbwayo A, Mutavi T, Weiner BJ, Collins P, Amanya C, Dorsey S. Applying human-centered design to maximize acceptability, feasibility, and usability of mobile technology supervision in Kenya: a mixed methods pilot study protocol. Implement Sci Commun. 2021 Jan 7;2(1):2. doi: 10.1186/s43058-020-00102-9. PMID 33413688
- [Derived] Dorsey S, Gray CL, Wasonga AI, Amanya C, Weiner BJ, Belden CM, Martin P, Meza RD, Weinhold AK, Soi C, Murray LK, Lucid L, Turner EL, Mildon R, Whetten K. Advancing successful implementation of task-shifted mental health care in low-resource settings (BASIC): protocol for a stepped wedge cluster randomized trial. BMC Psychiatry. 2020 Jan 8;20(1):10. doi: 10.1186/s12888-019-2364-4. PMID 31914959

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Children believed to be eligible were recruited using school enrollment lists, with the additional assistance of teachers and community health volunteers (CHVs) to confirm and locate them.
Pre-assignment Details: Due to the Stepped Wedge design, participants in Sequences 2-7 may have been screened twice: First, when their site served as a Comparison, and second, when their site was allocated to Intervention. Therefore, some children only contributed information at Comparison timepoints; if they were unavailable or ineligible when their site implemented, they were not randomized to receive the intervention via either delivery sector. Lost to follow-up refers to not completing the end-of-treatment survey.
Units Other Than Participants: Number of Sites
Groups:
- Sequence 1: March 26, 2018 - August 27, 2018 (Staggered delivery periods, with 8 once-per-week sessions per delivery period. Each site had separate girls and boys groups in both the health and education sector, for 4 total delivery periods in this sequence.)
- Sequence 2: January 28, 2019 - June 30, 2019 (Staggered delivery periods, with 8 once-per-week sessions per delivery period. Each site had separate girls and boys groups in both the health and education sector, for 4 total delivery periods in this sequence.)
- Sequence 3: May 6, 2019 - October 18, 2019 (Staggered delivery periods, with 8 once-per-week sessions per delivery period. Each site had separate girls and boys groups in both the health and education sector, for 4 total delivery periods in this sequence.)
- Sequence 4: January 27, 2020 - March 17, 2021 (Staggered delivery periods, with 8 once-per-week sessions per delivery period. Each site had separate girls and boys groups in both the health and education sector, for 4 total delivery periods in this sequence.)
  *Note: This Sequence experienced a prolonged hiatus due to the impact of COVID-19 on the school schedule in Kenya
- Sequence 5: January 28, 2021 - July 6, 2021 (Staggered delivery periods, with 8 once-per-week sessions per delivery period. Each site had separate girls and boys groups in both the health and education sector, for 4 total delivery periods in this sequence.)
  *Note: This Sequence was delayed due to the impact of COVID-19 on the school schedule in Kenya
- Sequence 6: May 27, 2021 - September 22, 2021 dates (Staggered delivery periods, with 8 once-per-week sessions per delivery period. Each site had separate girls and boys groups in both the health and education sector, for 4 total delivery periods in this sequence.)
  *Note: This Sequence was delayed due to the impact of COVID-19 on the school schedule in Kenya
- Sequence 7: October 27, 2021 - February 28, 2022 (Staggered delivery periods, with 8 once-per-week sessions per delivery period. Each site had separate girls and boys groups in both the health and education sector, for 4 total delivery periods in this sequence.)
  *Note: This Sequence was delayed due to the impact of COVID-19 on the school schedule in Kenya
Period: Overall Study
Arm/Group | Sequence 1 | Sequence 2 | Sequence 3 | Sequence 4 | Sequence 5 | Sequence 6 | Sequence 7
Started | 258; 10 Number of Sites | 151; 5 Number of Sites | 134; 5 Number of Sites | 127; 5 Number of Sites | 117; 5 Number of Sites | 85; 5 Number of Sites | 84; 5 Number of Sites
Completed | 256; 10 Number of Sites | 148; 5 Number of Sites | 119; 5 Number of Sites | 119; 5 Number of Sites | 116; 5 Number of Sites | 81; 5 Number of Sites | 75; 5 Number of Sites
Not Completed | 2; 0 Number of Sites | 3; 0 Number of Sites | 15; 0 Number of Sites | 8; 0 Number of Sites | 1; 0 Number of Sites | 4; 0 Number of Sites | 9; 0 Number of Sites
Not completed — Lost to Follow-up | 2 | 3 | 15 | 8 | 1 | 4 | 9

BASELINE CHARACTERISTICS:
Population: Participants with Baseline Characteristics data collected.
Groups:
- Youth Randomized to Health-Sector Delivered CBT: These child/adolescent participants and one of their guardians will receive Pamoja Tunaweza, the locally adapted version of Trauma-Focused Cognitive Behavioral Therapy, in a community setting from Community Health Volunteers.
  Trauma-Focused Cognitive Behavioral Therapy: Eight small-group sessions, including eight children and one guardian for each child, will meet separately, with joint activities in the final three sessions. TF-CBT will be delivered via community health volunteers in the community setting, and via selected teachers in the school setting--with two lay counselors leading the child group, and one leading the guardian group. Most TF-CBT components (psychoeducation, parenting, relaxation, cognitive coping, grief specific skills) will be delivered in groups, but 2-3 individual sessions mid-group will be used for imaginal exposure (i.e., talking about/processing traumatic events).
- Youth Randomized to Education-Sector Delivered CBT: These child/adolescent participants and one of their guardians will receive Pamoja Tunaweza, the locally adapted version of Trauma-Focused Cognitive Behavioral Therapy, in their school setting from teachers employed by their school.
  Trauma-Focused Cognitive Behavioral Therapy: Eight small-group sessions, including eight children and one guardian for each child, will meet separately, with joint activities in the final three sessions. TF-CBT will be delivered via community health volunteers in the community setting, and via selected teachers in the school setting--with two lay counselors leading the child group, and one leading the guardian group. Most TF-CBT components (psychoeducation, parenting, relaxation, cognitive coping, grief specific skills) will be delivered in groups, but 2-3 individual sessions mid-group will be used for imaginal exposure (i.e., talking about/processing traumatic events).
- Youth Who Were Not Randomized to Receive Pamoja Tunaweza CBT: These child/adolescent participants and one of their guardians did not receive Pamoja Tunaweza, the locally adapted version of Trauma-Focused Cognitive Behavioral Therapy.
- Total: Total of all reporting groups
Arm/Group | Youth Randomized to Health-Sector Delivered CBT | Youth Randomized to Education-Sector Delivered CBT | Youth Who Were Not Randomized to Receive Pamoja Tunaweza CBT | Total
Number analyzed (Participants) | 413 | 438 | 105 | 956
Age, Continuous [Mean (Standard Deviation); unit: years] | 12.4 (1.1) | 12.5 (1.1) | 13.1 (1.1) | 12.5 (1.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 197 | 221 | 66 | 484
  Male | 216 | 217 | 39 | 472
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 413 | 438 | 105 | 956
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 413 | 438 | 105 | 956
  White | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Kenya | 413 | 438 | 105 | 956

OUTCOME MEASURES:

1. Primary Outcome: Change in Posttraumatic Stress Symptoms (Child Report)
Description: Severity of posttraumatic stress symptoms, as assessed by the Child and Adolescent Trauma Screen (child report), including additional items validated locally. Higher scores represent more severe symptoms. The range of scores is 0 to 66. Scores are the sum of 22 items asking about how often specific things have bothered someone in the past 4 weeks. Each item is measured on a scale of 0 to 3, where 0=never happens and 3=almost always.
Time Frame: Baseline, End of 8-session Treatment (assessed up to 18 weeks)
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Youth Randomized to Health-Sector Delivered CBT | Youth Randomized to Education-Sector Delivered CBT | Youth Who Were Not Randomized to Receive Pamoja Tunaweza CBT
Number analyzed (Participants) | 413 | 438 | 105
score on a scale | -13.2 [-14.4 to -12.1] | -12.8 [-13.9 to -11.6] | -6.9 [-9.5 to -4.3]

2. Primary Outcome: Fidelity
Description: Ability of the group leader to adhere to established Trauma-Focused Cognitive Behavioral Therapy (TF-CBT) protocols and guidelines, as assessed by the Fidelity and Adherence Rating Scales developed by the study team. Assessed in each observed TF-CBT session by supervisors. Higher scores represent higher adherence to TF-CBT. Adherence is measured on a scale of 0 to 6. Scores reported are observations of Child groups.
Time Frame: End of first year of site implementation (2 groups, 8 sessions each)
Population: This is a site-level outcome. Teams of 3 counselors delivered the intervention in each site. They were observed and scored as a group-based observation.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Units Other Than Participants: Sites
Arm/Group | Health-Sector Delivered CBT | Education-Sector Delivered CBT
Number analyzed (Participants) | 407 | 433
Number analyzed (Sites) | 39 | 39
score on a scale | 4.1 [3.9 to 4.2] | 4.4 [4.3 to 4.6]

3. Primary Outcome: Number of Sites That Adopted the Intervention
Description: Adoption is a binary yes/no outcome defined as initiating and delivering the 8-session TF-CBT groups by a 3-counselor team and is measured by counselor self-report (and confirmed by supervisors who observed groups). Assessed for each "trimester" end for schools and communities, summarized over the year. We report the number of sites out of 40 total that adopted the intervention.
Time Frame: End of first year of site implementation (2 groups, 8 sessions each)
Population: This is a site level outcome indicating whether the 3-counselor team in each sector implemented the 8 sessions.
Measure: Count of Units; unit: Sites
Units Other Than Participants: Sites
Arm/Group | Health-Sector Delivered CBT | Education-Sector Delivered CBT
Number analyzed (Participants) | 413 | 438
Number analyzed (Sites) | 40 | 40
Sites | 40 | 40

4. Primary Outcome: Number of Sites That Sustained the Intervention
Description: Sustainment is a binary yes/no outcome defined as maintained delivery 2 years after the study intervention period (2 groups delivered within a calendar year, with at least 80% capacity as compared to their group enrollment during initial implementation). It is measured by counselor self-report (and confirmed by supervisors). At times the number of youth that would be 80% enrolled required rounding down to the nearest whole person. We report the number of sites out of 40 total that sustained the intervention.
Time Frame: Two years after the first TF-CBT groups for each site
Population: This is a site level outcome indicating whether the 3-counselor team in each sector maintained delivery 2 years after the study intervention period.
Measure: Count of Units; unit: Sites
Units Other Than Participants: Sites
Arm/Group | Health-Sector Delivered CBT | Education-Sector Delivered CBT
Number analyzed (Participants) | 413 | 438
Number analyzed (Sites) | 40 | 40
Sites | 16 | 10

5. Secondary Outcome: Change in Posttraumatic Stress Symptoms (Caregiver Report)
Description: Severity of posttraumatic stress symptoms, as assessed by the Child and Adolescent Trauma Screen (caregiver report), including additional items validated locally. Higher scores represent more severe symptoms. The range of scores is 0 to 66. Scores are the sum of 22 items asking about how often specific things have bothered someone in the past 4 weeks. Each item is measured on a scale of 0 to 3, where 0=never happens and 3=almost always.
Time Frame: Baseline, End of 8-session Treatment (assessed up to 18 weeks)
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Youth Randomized to Health-Sector Delivered CBT | Youth Randomized to Education-Sector Delivered CBT | Youth Who Were Not Randomized to Receive Pamoja Tunaweza CBT
Number analyzed (Participants) | 413 | 438 | 105
score on a scale | -17.1 [-18.3 to -16.0] | -17.1 [-18.3 to -16.0] | -8.4 [-11.9 to -5.0]

6. Secondary Outcome: Change in Depressive Symptoms (Child Report)
Description: Level of experienced depressive symptoms, as assessed by the Adolescent version of the Patient Health Questionnaire (8-question version) and additional items validated locally. Higher scores represent more severe symptoms. The range of scores is 0 to 36. Scores are the sum of 12 item asking how often items have bothered someone in the past 2 weeks. Each item is measured on a scale of 0 to 3, where 0=not at all happens and 3=nearly every day.
Time Frame: Baseline, End of 8-session Treatment (assessed up to 18 weeks)
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Youth Randomized to Health-Sector Delivered CBT | Youth Randomized to Education-Sector Delivered CBT | Youth Who Were Not Randomized to Receive Pamoja Tunaweza CBT
Number analyzed (Participants) | 413 | 438 | 105
score on a scale | -3.6 [-4.3 to -2.9] | -3.3 [-4.0 to -2.5] | -2.3 [-4.0 to -0.5]

7. Secondary Outcome: Change in Grief (Child Report)
Description: Level of grief related to a traumatic event experienced by the child, as assessed by the Inventory of Complex Grief. Higher scores represent more severe symptoms. The range of scores is 0 to 112. Scores are the sum of 28 items asking about how often they have experienced each item past month. Each item is measured on a scale of 0 to 4, where 0=almost never (less than once a month) and 4=always (several times a day).
Time Frame: Baseline, End of 8-session Treatment (assessed up to 18 weeks)
Measure: Mean (95% Confidence Interval); unit: score on a scale
Groups:
- Youth Randomized to Health-Sector Delivered CBT: Youth Randomized to Health-Sector Delivered CBT (Not to test Health-Sector delivery compared to Education-Sector delivered, but rather to ensure similar demographic variation between these two important sectors).
  These child/adolescent participants and one of their guardians will receive Pamoja Tunaweza, the locally adapted version of Trauma-Focused Cognitive Behavioral Therapy, in a community setting from Community Health Volunteers.
  Trauma-Focused Cognitive Behavioral Therapy: Eight small-group sessions, including eight children and one guardian for each child, will meet separately, with joint activities in the final three sessions. TF-CBT will be delivered via community health volunteers in the community setting, and via selected teachers in the school setting--with two lay counselors leading the child group, and one leading the guardian group. Most TF-CBT components (psychoeducation, parenting, relaxation, cognitive coping, grief specific skills) will be delivered in groups, but 2-3 individual sessions mid-group will be used for imaginal exposure (i.e., talking about/processing traumatic events).
- Youth Randomized to Education-Sector Delivered CBT: Youth Randomized to Education-Sector Delivered CBT (Not to test Health-Sector delivery compared to Education-Sector delivered, but rather to ensure similar demographic variation between these two important sectors.)
  These child/adolescent participants and one of their guardians will receive Pamoja Tunaweza, the locally adapted version of Trauma-Focused Cognitive Behavioral Therapy, in their school setting from teachers employed by their school.
  Trauma-Focused Cognitive Behavioral Therapy: Eight small-group sessions, including eight children and one guardian for each child, will meet separately, with joint activities in the final three sessions. TF-CBT will be delivered via community health volunteers in the community setting, and via selected teachers in the school setting--with two lay counselors leading the child group, and one leading the guardian group. Most TF-CBT components (psychoeducation, parenting, relaxation, cognitive coping, grief specific skills) will be delivered in groups, but 2-3 individual sessions mid-group will be used for imaginal exposure (i.e., talking about/processing traumatic events).
Arm/Group | Youth Randomized to Health-Sector Delivered CBT | Youth Randomized to Education-Sector Delivered CBT | Youth Who Were Not Randomized to Receive Pamoja Tunaweza CBT
Number analyzed (Participants) | 413 | 438 | 105
score on a scale | -23.0 [-24.9 to -21.0] | -22.9 [-25.0 to -20.8] | -10.8 [-16.1 to -5.5]

8. Secondary Outcome: TF-CBT Knowledge Score
Description: Test of the level of knowledge of the lay counselors about TF-CBT, as assessed by the TF-CBT Knowledge Assessment. Higher scores represent greater group leader knowledge of TF-CBT. Scores could range from 0 to 32.5. The knowledge test was administered to all lay counselors at the end of their TF-CBT training to confirm their readiness to deliver the intervention. For each sequence, training occurred just before implementation of the intervention.
Time Frame: Immediately Post-Training (on final day of training for the sequence, up to 6 days)
Population: This is a group leader-level outcome.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Units Other Than Participants: Group Leaders
Arm/Group | Health-Sector Delivered CBT | Education-Sector Delivered CBT
Number analyzed (Participants) | 413 | 438
Number analyzed (Group Leaders) | 97 | 104
score on a scale | 25.1 [24.4 to 25.8] | 27.8 [27.1 to 28.4]

9. Secondary Outcome: Change in Prosocial Behavior (Child Report)
Description: Change in behavioral strengths of the child, as assessed by the Prosocial Behavior subscale of the Strengths and Difficulties Questionnaire before and after the intervention. There are 5 items asking about the degree to which the child reports prosocial behavior. Each item has 3 possible responses on a scale of 0 to 2, where 0=not at all true and 2=certainly true. The total score summing across the 5 items could range from 0 to 10. Higher scores are more favorable, representing more prosocial behavior.
Time Frame: Baseline, End of 8-session Treatment (assessed up to 18 weeks)
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Youth Randomized to Health-Sector Delivered CBT | Youth Randomized to Education-Sector Delivered CBT | Youth Who Were Not Randomized to Receive Pamoja Tunaweza CBT
Number analyzed (Participants) | 413 | 438 | 105
score on a scale | 0.09 [-0.1 to 0.3] | 0.2 [0.03 to 0.4] | 0.2 [-0.2 to 0.6]

10. Secondary Outcome: Change in Behavioral Problems (Guardian Report)
Description: Change in behavioral problems of the child, as assessed by the Conduct Problems subscale of the Strengths and Difficulties Questionnaire, including additional items validated locally. There are 9 items asking about the degree to which the guardian reports conduct problems observed in the child. Each item has 3 possible responses on a scale of 0 to 2, where 0=not at all true and 2=certainly true. The total score summing across the 5 items could range from 0 to 18. Lower scores are more favorable, representing decreased behavioral problems.
Time Frame: Baseline, End of 8-session Treatment (assessed up to 18 weeks)
Measure: Mean (95% Confidence Interval); unit: score on a scale
Groups:
- Youth Randomized to Health-Sector Delivered CBT: Youth Randomized to Health-Sector Delivered CBT (Not to test Health-Sector delivery compared to Education-Sector delivered, but rather to ensure similar demographic variation between these two important sectors.)
  These child/adolescent participants and one of their guardians will receive Pamoja Tunaweza, the locally adapted version of Trauma-Focused Cognitive Behavioral Therapy, in a community setting from Community Health Volunteers.
  Trauma-Focused Cognitive Behavioral Therapy: Eight small-group sessions, including eight children and one guardian for each child, will meet separately, with joint activities in the final three sessions. TF-CBT will be delivered via community health volunteers in the community setting, and via selected teachers in the school setting--with two lay counselors leading the child group, and one leading the guardian group. Most TF-CBT components (psychoeducation, parenting, relaxation, cognitive coping, grief specific skills) will be delivered in groups, but 2-3 individual sessions mid-group will be used for imaginal exposure (i.e., talking about/processing traumatic events).
Arm/Group | Youth Randomized to Health-Sector Delivered CBT | Youth Randomized to Education-Sector Delivered CBT | Youth Who Were Not Randomized to Receive Pamoja Tunaweza CBT
Number analyzed (Participants) | 413 | 438 | 105
score on a scale | -0.9 [-1.1 to -0.7] | -0.7 [-0.9 to -0.5] | -0.04 [-0.5 to 0.6]

11. Secondary Outcome: School Attendance
Description: School attendance measured by the number of school days missed in the past two weeks, as reported by the guardian.
Time Frame: Baseline
Measure: Mean (95% Confidence Interval); unit: days
Arm/Group | Youth Randomized to Health-Sector Delivered CBT | Youth Randomized to Education-Sector Delivered CBT | Youth Who Were Not Randomized to Receive Pamoja Tunaweza CBT
Number analyzed (Participants) | 413 | 438 | 105
days | 2.1 [1.8 to 2.4] | 1.9 [1.6 to 2.2] | 1.1 [0.7 to 1.5]

12. Secondary Outcome: Change in Proportion of Children Engaged in Excessive Child Labor for Pay
Description: Change in proportion of children engaged in excessive child labor for pay in the past week, as assessed by the Child Work and Labor Questionnaire and reported by the child. UNICEF's definition of excessive labor for children aged 12 and older is 14 hours per week for pay and 28 hours per week with or without pay. This is constructed as a binary variable, and we present a difference in the proportion of children who worked 14 or more hours in the past week for income-generating activities (work without pay was not assessed). Lower proportion is more favorable, representing fewer children engaged in excessive child labor for pay.
Time Frame: Baseline to third annual follow-up
Population: Participants who were assessed at the third annual follow-up and were at least 16 years old at follow-up time.
Measure: Mean (95% Confidence Interval); unit: proportion of youth
Arm/Group | Youth Randomized to Health-Sector Delivered CBT | Youth Randomized to Education-Sector Delivered CBT | Youth Who Were Not Randomized to Receive Pamoja Tunaweza CBT
Number analyzed (Participants) | 129 | 142 | 25
proportion of youth | 0.1 [0.05 to 0.2] | 0.09 [0.03 to 0.2] | 0.12 [0.01 to 0.3]

13. Secondary Outcome: Change in Proportion of Children Engages in Excessive Household Assistance Without Pay
Description: Change in proportion of children engaged in chores (non-income generating work around the home) in the past week, as reported by the child. This is constructed as a binary variable, and we present a difference in the proportion of children who did chores for 14 or more hours in the past week. Lower proportion is more favorable, representing fewer children engaged in excessive household assistance without pay.
Time Frame: Baseline to third annual follow-up
Population: Participants who were assessed at the third annual follow-up and were at least 16 years old at follow-up time.
Measure: Mean (95% Confidence Interval); unit: proportion of youth
Arm/Group | Youth Randomized to Health-Sector Delivered CBT | Youth Randomized to Education-Sector Delivered CBT | Youth Who Were Not Randomized to Receive Pamoja Tunaweza CBT
Number analyzed (Participants) | 129 | 142 | 25
proportion of youth | 0.3 [0.2 to 0.5] | 0.3 [0.2 to 0.4] | 0.2 [-0.07 to 0.6]

14. Secondary Outcome: Safer Sex Peer Norms Score
Description: Agreement exhibited by the child with positive peer norms regarding sexual behavior, as assessed by the Safer Sex Peer Norms subscale on the Safer Sex Peer Norms and Substance Use Questionnaire. This measure is only administered if the child is 16 or older, so for this outcome, we report specifically on the Safer Sex Peer Norms assessment collected at the 3rd annual follow-up timepoint. Scores are the sum of 7-item asking about agreement with the item. Each item is measured on a scale of 1 to 4, where 1=strongly disagree and 4=strongly agree. The range of total scores is 0 to 28. Higher scores are more favorable, representing stronger agreement with positive peer norms.
Time Frame: Third annual follow-up
Population: Participants who were assessed at the third annual follow-up and were at least 16 years old at follow-up time.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Youth Randomized to Health-Sector Delivered CBT | Youth Randomized to Education-Sector Delivered CBT | Youth Who Were Not Randomized to Receive Pamoja Tunaweza CBT
Number analyzed (Participants) | 124 | 137 | 23
score on a scale | 16.3 [15.6 to 17.1] | 16.7 [16.0 to 17.4] | 16.5 [14.9 to 18.1]

15. Secondary Outcome: Change in Proportion of Children Reporting Any Current Substance Use
Description: Change in proportion of children reporting any current alcohol, tobacco, or other drug use, as assessed by the Safer Sex Peer Norms and Substance Use Questionnaire and reported by the child. This is reported as a binary variable representing the proportion of children who report current drug use or drinking alcohol in the past 7 days or using tobacco in the past 7 days. Lower proportion is more favorable.
Time Frame: Baseline to third annual follow-up
Population: Participants who were assessed at the third annual follow-up and were at least 16 years old at follow-up time.
Measure: Mean (95% Confidence Interval); unit: proportion of youth
Arm/Group | Youth Randomized to Health-Sector Delivered CBT | Youth Randomized to Education-Sector Delivered CBT | Youth Who Were Not Randomized to Receive Pamoja Tunaweza CBT
Number analyzed (Participants) | 129 | 142 | 25
proportion of youth | -0.01 [-0.05 to 0.02] | -0.02 [-0.03 to 0.01] | 0.0 [0.0 to 0.0]

16. Other Pre Specified Outcome: Relationship Closeness
Description: Closeness of the child's relationship with their caregiver, as assessed by caregiver report in the Closeness subscale of the Child-Parent Relationship Scale. Higher scores represent greater closeness.
Time Frame: End of 8-session Treatment (assessed up to 18 weeks)
Reporting Status: Not Posted

17. Other Pre Specified Outcome: Relationship Conflict
Description: Conflict in the child's relationship with their caregiver, as assessed by caregiver report in the Conflict subscale of the Child-Parent Relationship Scale. Higher scores represent more conflict.
Time Frame: End of 8-session Treatment (assessed up to 18 weeks)
Reporting Status: Not Posted

18. Other Pre Specified Outcome: Guardian-provided Social Support
Description: Social support provided to the child by their parent or guardian, as assessed by child report in the Child and Adolescent Social Support Scale. Higher scores represent more support.
Time Frame: End of 8-session Treatment (assessed up to 18 weeks)
Reporting Status: Not Posted

19. Other Pre Specified Outcome: Intervention Acceptability
Description: Assessed using both reflective and formative measures at the group leader level. The reflective measure is the Acceptability of Intervention Measure (AIM), with scores ranging from 1 (least acceptable) to 5 (most acceptable) calculated as a mean score to reflect the acceptability of the TF-CBT intervention in a given setting. The formative measure is the Johns Hopkins University (JHU) Implementation science case for Acceptability (using only 5 items that mapped directly onto Proctor's definition of acceptability and did not overlap with items on the AIM measure). This is not treated as a scale, and items are analyzed independently of each other.
Time Frame: End of first year of site implementation (2 groups, 8 sessions each)
Reporting Status: Not Posted

20. Other Pre Specified Outcome: Intervention Feasibility
Description: Assessed using both reflective and formative measures at the group leader level. The reflective measure is the Feasibility of Intervention Measure (FIM), with scores ranging from 1 (least feasible) to 5 (most feasible) calculated as a mean score to reflect the feasibility of implementing TF-CBT in a given setting. The formative measure is the Johns Hopkins University Implementation science scale for Feasibility (using 12 items). This is not treated as a scale, and items are analyzed independently of each other. 2 additional items were included that inquired about the estimated hours per week that respondents felt Pamoja Tunaweza/TF-CBT would require, given the importance of this information for understanding added workload and feasibility for providers in the two contexts ("On average, how many hours per week do you spend on Pamoja Tunaweza/TF-CBT [e.g., preparing for sessions, delivering sessions, and supervision]?").
Time Frame: End of first year of site implementation (2 groups, 8 sessions each)
Reporting Status: Not Posted

21. Other Pre Specified Outcome: Intervention Appropriateness
Description: A formative measure is used to assess perceived appropriateness of the TF-CBT intervention at the group leader level, with scores ranging from 1 (least appropriate) to 5 (most appropriate). This is not treated as a scale, and items are analyzed independently of each other. Six items were adapted from the Johns Hopkins University implementation measures that aligned with Proctor and colleagues' (20) definition of appropriateness. Minor changes were made to fit wording to the local context. Two additional items were developed to measure appropriateness domain content for which Johns Hopkins University items did not exist. Given challenges in creating new items, Hujig's Theoretical Domains Framework was used when possible to guide item creation (42). In the resulting 8-item measure, 4 items assessed the perceived fit of delivering TF-CBT with one's role. The additional 4 items assessed the perceived fit of delivering TF-CBT within the specific setting.
Time Frame: End of first year of site implementation (2 groups, 8 sessions each)
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Enrollment through final annual follow-up assessment (maximum three years post-intervention, depending on stepped-wedge sequence timing)
Groups:
- Youth Randomized to Health-Sector Delivered CBT: These child/adolescent participants and one of their guardians received Pamoja Tunaweza, the locally adapted version of Trauma-Focused Cognitive Behavioral Therapy, in a community setting from Community Health Volunteers.
  Trauma-Focused Cognitive Behavioral Therapy: Eight small-group sessions, including eight children and one guardian for each child, will meet separately, with joint activities in the final three sessions. TF-CBT will be delivered via community health volunteers in the community setting, and via selected teachers in the school setting--with two lay counselors leading the child group, and one leading the guardian group. Most TF-CBT components (psychoeducation, parenting, relaxation, cognitive coping, grief specific skills) will be delivered in groups, but 2-3 individual sessions mid-group will be used for imaginal exposure (i.e., talking about/processing traumatic events).
- Youth Randomized to Education-Sector Delivered CBT: These child/adolescent participants and one of their guardians received Pamoja Tunaweza, the locally adapted version of Trauma-Focused Cognitive Behavioral Therapy, in their school setting from teachers employed by their school.
  Trauma-Focused Cognitive Behavioral Therapy: Eight small-group sessions, including eight children and one guardian for each child, will meet separately, with joint activities in the final three sessions. TF-CBT will be delivered via community health volunteers in the community setting, and via selected teachers in the school setting--with two lay counselors leading the child group, and one leading the guardian group. Most TF-CBT components (psychoeducation, parenting, relaxation, cognitive coping, grief specific skills) will be delivered in groups, but 2-3 individual sessions mid-group will be used for imaginal exposure (i.e., talking about/processing traumatic events).
- Youth Who Did Not Receive Pamoja Tunaweza CBT: These child/adolescent participants and one of their guardians did not receive Pamoja Tunaweza, the locally adapted version of Trauma-Focused Cognitive Behavioral Therapy.
Arm/Group | Youth Randomized to Health-Sector Delivered CBT | Youth Randomized to Education-Sector Delivered CBT | Youth Who Did Not Receive Pamoja Tunaweza CBT
All-Cause Mortality (participants affected / at risk) | 0/413 | 0/438 | 0/105
Serious Adverse Events (participants affected / at risk) | 0/413 | 0/438 | 0/105
Other Adverse Events (participants affected / at risk) | 0/413 | 0/438 | 0/105

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-01-08): https://cdn.clinicaltrials.gov/large-docs/96/NCT03243396/Prot_SAP_000.pdf
  • Informed Consent Form (2021-05-06): https://cdn.clinicaltrials.gov/large-docs/96/NCT03243396/ICF_001.pdf